CLINICAL TRIAL: NCT02160665
Title: A Double-Blind,Randomized,Parallel-Group,Vehicle-Controlled,Multi-Center Study Comparing a Generic Tazarotene Cream, 0.05% to RLD Tazorac® Cream, 0.05% and Both Treatments to a Vehicle in the Treatment of Plaque Psoriasis
Brief Title: Generic Tazarotene Cream, 0.05% for the Treatment of Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: G & W Laboratories Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SYM 2013-01
Record Dates: First submitted 2014-06-09; First posted 2014-06-11 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — tazarotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vehicle (Placebo Comparator): Vehicle of Test product (G & W Laboratories, Inc.)
  Interventions: Drug: Vehicle
- Reference: Tazorac Cream, 0.05% (Other): Reference: Tazorac (tazarotene) Cream, 0.05% (Allergan, Inc.)
  Interventions: Drug: Reference: Tazorac Cream, 0.05%
- Test:Tazarotene Cream, 0.05% (Active Comparator): Test: Tazarotene Cream, 0.05% (G & W Laboratories, Inc.)
  Interventions: Drug: Tazarotene Cream, 0.05%

INTERVENTIONS:
Drug: Tazarotene Cream, 0.05% — Tazarotene Cream, 0.05% (G & W Laboratories, Inc.)
  Other Names: Test
  Arms: Test:Tazarotene Cream, 0.05%
Drug: Vehicle — Vehicle of Test product (G & W Laboratories, Inc.)
  Other Names: Placebo
  Arms: Vehicle
Drug: Reference: Tazorac Cream, 0.05% — Reference: Tazorac (tazarotene) Cream, 0.05% (Allergan, Inc.)
  Other Names: Tazorac
  Arms: Reference: Tazorac Cream, 0.05%

SUMMARY:
The purpose of this study is to compare the safety and efficacy profiles of Tazarotene Cream, 0.05% and Tazorac® (Tazarotene) Cream, 0.05% in order to demonstrate bioequivalence and to demonstrate the superiority of the 2 active creams over that of the Vehicle (placebo) in the treatment of plaque psoriasis.

DETAILED DESCRIPTION:
This is a double-blind, randomized, parallel-group, vehicle-controlled, multicenter study of Tazarotene Cream, 0.05% in subjects with plaque psoriasis. Subjects will be randomly assigned in a 1:1:1 ratio to Test, Reference, or Vehicle.

Subjects will be admitted into the study after informed consent has been obtained and all inclusion/exclusion criteria have been met. At each visit, the same investigator (whenever possible) will grade the clinical signs of plaque psoriasis at the designated target lesion site using the Psoriasis Area Severity Index (PASI), an Investigator's Global Assessment (IGA) of disease severity will be performed (IGA scores range from 0 = none to 5 = very severe), and application site reactions (erythema, dryness, burning/stinging, erosion, edema, pain, and pruritus) will be assessed. In addition, the involved body surface area (BSA) will be determined at Visit 1 and Visit 4. Safety will be assessed by monitoring all adverse events (AEs) at each visit and a telephone contact at Day 7 (+ 4 days)

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the study
2. Be male or female, at least 18 years of age
3. Have a definite clinical diagnosis of stable (at least 6 months) plaque psoriasis, involving at least 2% and no more than 20% of the body surface area (BSA) (not including the scalp and intertriginous areas)
4. Have a minimum plaque elevation at the target lesion site of at least moderate severity (grade ≥ 3 on the Psoriasis Area Severity Index [PASI]). The most severe lesion at baseline should be identified as the target lesion
5. Have an Investigator's Global Assessment (IGA) of disease severity of at least moderate (score ≥ 3) as an overall assessment of all lesions to be treated.
6. Be in general good health and free from any clinically significant disease other than psoriasis that might interfere with the study evaluations
7. Be willing and able to understand and comply with the requirements of the study, apply the study medication as instructed, return for the required treatment period visits, comply with therapy prohibitions, and be able to complete the study
8. Female subjects of childbearing potential (excluding women who are surgically sterilized or postmenopausal for at least 2 years) must have a negative urine pregnancy test having sensitivity down to at least 50 mIU/ml for hCG, begin treatment during a normal menstrual period and must be willing to use an acceptable method of contraception during the study. The following are considered acceptable methods of birth control for the purpose of this study: oral contraceptives, contraceptive patches, contraceptive implant, vaginal contraceptive, double barrier methods (e.g., condom and spermicide), contraceptive injection (Depo-Provera®), intrauterine device (IUD), hormonal IUD (Mirena®), and abstinence with a documented second acceptable method of birth control if the subject becomes sexually active. Subjects entering the study who are on hormonal contraceptives must have been on the method for at least 90 days prior to the study and continue the method for the duration of the study. Subjects who had used hormonal contraception and stopped must have stopped no less than 90 days prior to Visit 1/Day 1
9. Be willing to limit sun exposure overall, maintain a reasonably constant exposure, and avoid use of tanning booths or other UV light sources during their participation in the study

Exclusion Criteria:

1. A female subject who is pregnant, nursing, planning a pregnancy, or does not agree to use an acceptable form of birth control within the study participation period
2. Have a current diagnosis of unstable forms of psoriasis in the treatment area, including pustular, guttate, exfoliative or erythrodermic psoriasis
3. Have a history of psoriasis unresponsive to topical treatments
4. Have other inflammatory skin disease in the treatment area that may confound with the evaluation of plaque psoriasis (e.g., atopic dermatitis, contact dermatitis, eczema, tinea corporis)
5. Have pigmentation, extensive scarring, pigmented lesions, or sunburn in the treatment areas that could interfere with the rating of efficacy parameters
6. Have an unstable medical disorder, life-threatening disease, or current malignancy
7. Have current immunosuppression
8. Have received any treatment listed in Table 8 1 more recently than the indicated washout period prior to Visit 1/Day 1
9. Would continue to receive any treatment listed in Table 8 1 during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 866 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
primary efficacy endpoint | Week 12
  The primary efficacy endpoint is the proportion of subjects with treatment success on the IGA at Visit 4/Week 12. Treatment success is defined as absent, very mild, or mild disease shown by a score of 0, 1, or 2 within the treatment area on the IGA. The primary analyses include evaluation of bioequivalence between the 2 active products and evaluations of superiority of each active treatment over the vehicle.

SECONDARY OUTCOMES:
Proportion of subjects with disease severity | Week 12
  Secondary efficacy endpoints will include: 1) the proportion of subjects with disease severity at Visit 4/Week 12 consistent with absent or very mild disease shown by a score of 0 or 1 within the treatment area on the IGA
the proportion of subjects with target lesion site | Week 12
  the proportion of subjects with target lesion site plaque elevation, scaling, and erythema scores of ≤ 1 on the PASI at Visit 4/Week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bukhalo, MD, Principal Investigator — Altman Dermatology Associates
Locations (1):
- Altman Dermatology Associates, Arlington Heights, Illinois, United States

IPD SHARING:
Plan to Share IPD: No